CLINICAL TRIAL: NCT03402113
Title: The Effect of Different Sedation Protocols on Skeletal Muscle Metabolism in Mechanical Ventilated Patients
Brief Title: Sedation Protocols and Skeletal Muscle Metabolism in Mechanical Ventilated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gulou ICU
Record Dates: First submitted 2017-12-26; First posted 2018-01-18 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2017-12

CONDITIONS: Hypercatabolism; Sedative, Hypnotic, or Anxiolytic Use Disorders
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine consistent infusion as sedative.
  Interventions: Drug: Dexmedetomidine
- Midazolam group (Active Comparator): Midazolam consistent infusion as sedative.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — consistent infusion at a loading dose of 0.15ug/kg/h, increased by 0.15ug/kg/h, with a maximum dose of 1.5ug/kg/h.
  Arms: Dexmedetomidine group
Drug: Midazolam — consistent infusion at a loading dose of 1mg/h, increased by 1mg/h, with a maximum dose of 10mg/h.
  Arms: Midazolam group

SUMMARY:
To investigate the effects of different sedation protocols on skeletal muscle metabolism in mechanical ventilated patients in ICU. Mechanical ventilated patients who are anticipated to stay in ICU for more than 5 days are enrolled and randomly assigned to the following three groups, interventional group(dexmedetomidine), control group(midazolam) and no sedation group. Serum, CT scan of intercostal muscles, ultrasound evaluation of quadriceps femoris are obtained.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilated for more than 48h
* 18-80 years
* stay in ICU for more than 5 days

Exclusion Criteria

* already participated in other clinical trials
* pregnancy or lactation
* lower limb amputation
* primary neuro-muscular disease
* disseminated tumor or accepted special therapy
* alcohol abuse
* severe liver dysfunction(Child-Push C)
* unstable angina/acute myocardial infarction
* heart rates<50bpm
* all kinds dialysis
* severe burn
* epidural anesthesia
* severe neurological disease（acute stroke, uncontrollable epilepsy, severe dementia, etc）

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
acute muscle wasting | From date of randomization to extubation,up to 7 days
  measured by 3-MH release in serum

SECONDARY OUTCOMES:
28-day mortality | From date of randomization to date of death from any cause,up to 28 days
  death rate within 28 days after mechanical ventilation
length of ICU stay | From date of randomization to date of to discharge or death,up to 28 days
  time from enrollment to discharge or die

CONTACTS AND LOCATIONS:
Locations (1):
- The Affliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not available to other researchers after publication.